CLINICAL TRIAL: NCT00735345
Title: Chemotherapy Induction and Chemoradiotherapy Combined With Cetuximab Respectively in Patients With Non-Metastatic Esophageal Carcinoma: A Multicentric Phase II Study
Brief Title: Chemotherapy Induction and Chemoradiotherapy in Patients With Esophageal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: because of safety concerns the study was terminated prematurely
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry)
Responsible Party: Prof. Dr. Richard Greil, Arbeitsgemeinschaft medikamentoese Tumortherapie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_ECa; EudraCT Nr. 2008-001016-21
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Pre-operative; Chemo-immunotherapy; Radiochemo-immunotherapy; EGFR; Radiosensitivity; Resection
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorouracil; Cisplatin; Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Chemo induction therapy followed by chemoradiotherapy and surgical resection or definitive radiotherapy
  Interventions: Drug: 5-FU; Drug: Cisplatin; Drug: Taxotere; Biological: Cetuximab; Radiation: Radiation during chemoradio-immunotherapy

INTERVENTIONS:
Drug: 5-FU — 750 mg/m2/d C.I. i.v.d1-5, d29-33 and 300 mg/m2/d C.I. i.v. on the days of radiotherapy
Drug: Cisplatin — 15 mg/m2/d i.v. d1-5, d29-33
Drug: Taxotere — 75 mg/m2/d i.v. d1 and d29, 15 mg/m2/d i.v. on d57, d64, d71 and d78
  Other Names: Docetaxel
Biological: Cetuximab — Cetuximab: 400 mg/m2 i.v. d1; 250mg/m2 weekly d8 through d85
  Other Names: Erbitux
Radiation: Radiation during chemoradio-immunotherapy — 39.6 Gy total dose

SUMMARY:
The aim of this study is the evaluate the feasibility and safety of chemotherapy induction treatment combined with cetuximab followed by chemoradiotherapy combined with cetuximab in the treatment of patients with non-metastatic esophageal cancer.

DETAILED DESCRIPTION:
Patients with a locoregional carcinoma of the esophagus or gastro-esophageal junction have a low survival prognosis following surgical resection. In studies published to date no positive effect upon overall survival could be demonstrated for preoperative chemotherapy or chemoradiotherapy. However, patients with a complete remission following preoperative therapy show prolonged survival.

This study design is based upon decreasing primary tumour and preventing oder delaying micrometastases by means of a chemo induction therapy, increasing R0 resection rates and preventing local recurrence by means of preoperative chemoradiotherapy, increasing the radiosensitivity of tumour cells through treatment combination with cetuximab, surgical resection of the locoregional primary tumour or definitive radiochemotherapy in case the primary tumour is inoperable.

The aim of this study is therefore to evaluate the feasibility and safety of a 3-staged therapy approach including an EGFR antibody in the treatment of patients with potentially resectable esophageal cancer, as well as the evaluation of objective response rates to this preoperative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* histologically confirmed esophageal cancer (squamous cell carcinoma)
* measurable, non-metastatic disease (uT1-4)
* no previous cancer therapy (chemotherapy, radiotherapy or resection)
* life expectancy > 3 months
* age > 18 years
* WHO Status ≤ 2
* negative pregnancy test for women of child-bearing potential, and use of adequate contraception
* hematological status: neutrophiles ≥ 1,5x10E9/L, thrombocytes ≥ 100x10E9/L
* adequate renal function: serum creatinine ≤ 1,5 x ULN
* adequate liver function: alkaline phosphatase < 2,5 x ULN, total bilirubin < 1,5 x ULN

Exclusion Criteria:

* pregnant or nursing women
* women of child-bearing potential without adequate contraception
* concomitant anti-tumoral therapy except study mandated procedures
* cervical esophageal cancer or diagnosis of metastases
* participation in other clinical trials within the last 30 days
* history of malignant disease within the last 5 years
* peripheral neuropathy (NCI CTC ≥ grade 1)
* concurrent active and serious non-malignant diseases: uncontrolled heart insufficiency, angina pectoris, hypertension or arrhythmias, liver disease, significant neurological or psychiatric conditions
* active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response rate | Duration of study
Percentage of complete remissions and resection rate | Duration of study

SECONDARY OUTCOMES:
Occurrence of toxicities | Duration of study
Evaluation of Quality of Life | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Eisterer, Prof. Dr., Principal Investigator — Medizinische Universitaet Innsbruck
Locations (7):
- Austria (7):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Universitätsklinikum Graz, Graz
  - Universitätsklinik Innsbruck, Innsbruck
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus Barmherzige Brueder St. Veit a.d. Glan, Saint Veit/ Glan
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - Klinikum Kreuzschwestern Wels GmbH, Wels